CLINICAL TRIAL: NCT00144911
Title: A Randomized, Double-Blind, Parallel Group, 52-Week Study to Compare the Effect of Fluticasone Propionate/Salmeterol DISKUS® Inhaler Combination Product 250/50mcg Twice Daily With Salmeterol DISKUS® Inhaler 50mcg Twice Daily on the Annual Rate of Moderate/Severe Exacerbations in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: ADVAIR® DISKUS® Inhaler (Fluticasone Propionate/Salmeterol) Versus SEREVENT® DISKUS® Inhaler (Salmeterol) For The Treatment Of Chronic Obstructive Pulmonary Disease Exacerbations. ADVAIR® DISKUS® Inhaler and SEREVENT® DISKUS® Inhaler Are Trademarks of the GSK Group of Companies.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCO40043
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: exacerbations; breathing; chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration | interventions — Salmeterol Xinafoate; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Salmeterol; Drug: Fluticasone Propionate/Salmeterol Combination Product

INTERVENTIONS:
Drug: Salmeterol
Drug: Fluticasone Propionate/Salmeterol Combination Product
  Other Names: Salmeterol

SUMMARY:
This study evaluates the effect of two medicines on COPD (Chronic Obstructive Pulmonary Disease) exacerbations. This study will last up to 56 weeks, and subjects will visit the clinic 10 times. Subjects will be given breathing tests and will record their breathing symptoms daily on diary cards. All study related medicines and medical examinations will be provided at no cost. The two drugs used in this study have been approved by the FDA for use in patients with COPD.

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Parallel Group, 52-week Study to Compare the Effect of the Fluticasone Propionate/Salmeterol DISKUS® inhaler Combination Product 250/50mcg twice daily (BID) with Salmeterol DISKUS® inhaler 50mcg BID on the Annual Rate of Moderate/Severe Exacerbations in Subjects with Chronic Obstructive Pulmonary Disease (COPD)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD (chronic obstructive pulmonary disease).
* Current or previous cigarette smokers with a smoking history of at least 10 pack-years.
* History of a least 1 COPD exacerbation in the 12 months prior to screening.
* Forced expiratory volume in one second (FEV1) of less than or equal to 50% of predicted normal.

Exclusion Criteria:

* Current diagnosis of asthma.
* Additional respiratory disorders other than COPD (eg, sarcoidosis, alpha-1 antitrypsin deficiency, cystic fibrosis, or active tuberculosis).
* Concurrent use of long-acting beta-agonists, long-acting anticholinergics, inhaled and oral corticosteroids, theophylline, investigational medications, ritonavir, and anti-leukotrienes.
* Lung resection surgery within 1 year of screening.
* Abnormal and clinically significant ECG findings at screening.
* Other inclusion and exclusion criteria will be evaluated at the first study visit.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Actual)
Dates: Start 2004-10; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Rate of moderate/severe exacerbations over a 52 week treatment period.

SECONDARY OUTCOMES:
The time until the first moderate/severe exacerbation, the annual rate of exacerbations requiring oral corticosteroid treatment, and breathing tests conducted over one year.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (93):
- United States (81):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Corona, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Palmdale, California
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, Rancho Mirage, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Sepulveda, California
  - GSK Investigational Site, Stockton, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Englewood, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Largo, Florida
  - GSK Investigational Site, North Miami Beach, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Champaign, Illinois
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Des Moines, Iowa
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, Slidell, Louisiana
  - GSK Investigational Site, Auburn, Maine
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Cherry Hill, New Jersey
  - GSK Investigational Site, Summit, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Larchmont, New York
  - GSK Investigational Site, Lewistown, New York
  - GSK Investigational Site, Elizabeth City, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Statesville, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Cumberland, Rhode Island
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, Corsicana, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Abingdon, Virginia
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Newport News, Virginia
  - GSK Investigational Site, Gig Harbor, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Morgantown, West Virginia
- Canada (12):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Grimsby, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Cowansville, Quebec
  - GSK Investigational Site, La Malbaie, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Saint-Léonard, Quebec
  - GSK Investigational Site, Sainte Jerome, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Sorel-Tracy, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Ferguson GT, Anzueto A, Fei R, Emmett A, Knobil K, Kalberg C. Effect of fluticasone propionate/salmeterol (250/50 microg) or salmeterol (50 microg) on COPD exacerbations. Respir Med. 2008 Aug;102(8):1099-108. doi: 10.1016/j.rmed.2008.04.019. Epub 2008 Jul 9. PMID 18614347
- [Derived] Disantostefano RL, Li H, Rubin DB, Stempel DA. Which patients with chronic obstructive pulmonary disease benefit from the addition of an inhaled corticosteroid to their bronchodilator? A cluster analysis. BMJ Open. 2013 Apr 22;3(4):e001838. doi: 10.1136/bmjopen-2012-001838. Print 2013. PMID 23613569
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: SCO40043 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SCO40043 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SCO40043 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SCO40043 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SCO40043 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SCO40043 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SCO40043 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register